CLINICAL TRIAL: NCT03841578
Title: Effects of Dark Chocolate on Gastrointestinal Motility in Healthy Subjects
Brief Title: Dark Chocolate and Intestinal Motility
Acronym: CHOCO-mot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, PhD MD Professor Piero Portincasa, University of Bari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1519UO
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Gastrointestinal Motility
Keywords: Dark chocolate, gastrointestinal motility

STUDY DESIGN:
Intervention Model Description: 10 healthy subjects (controls) undergoing organoleptic assessment and gastrointestinal motility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy (Experimental): 10 participants (matched per gender), aged 25-35 years old who accepts the consumption of dark chocolate plus a 'NutriDrink' previous to signing an informed consent and providing authorization to the handling of their personal data
  Interventions: Dietary Supplement: Healthy

INTERVENTIONS:
Dietary Supplement: Healthy — 25g of dark chocolate (70%) will be provided to participants on Phase 1 (organoleptic assessment). On Phase 2 (gastrointestinal motility assessment), they will ingest a standard liquid meal (NutriDrink, 200ml), consisting of 10g of lactulose and 12g of fat

SUMMARY:
Following food intake, the body activates several processes to degrade and digest it. Studies show that there is an adaptation of gastric emptying and gastrointestinal motility to a food component; therefore, considering the intestinal adaptation to chocolate, the effect on gastrointestinal motility in relation to the intake of chocolate will be investigated.

The organoleptic perceptions of dark chocolate will also be analyzed to evaluate the appreciation of the product ingested by the subject.

DETAILED DESCRIPTION:
Chocolate, the main product deriving from cocoa beans (Theobroma cacao, from the Greek "food of the gods") has its origin in Mexico, where Maya, Inca and Aztecs practiced its cultivation, has for centuries been appreciated for its pleasant taste and its beneficial health effects.

Chocolate is the most sought-after food worldwide, and currently its consumption has increased considerably with a wide availability of products on the market.

Dietary choices are strongly influenced by the taste and consistency of foods. Fat is largely responsible for the sensory properties of many foods and, therefore, contribute greatly to the pleasure of eating. Dark chocolate consists of ≈43% of lipids, mainly represented by cocoa butter. Cocoa butter is composed of an average of 33% of oleic acid, 25% of palmitic acid and 33% of stearic acid. Another component of chocolate is polyphenols, in particular flavonoids, substances with numerous beneficial effects for health, including antihypertensive, anti-inflammatory, antithrombotic, metabolic and prebiotic activity playing a role in the change of human intestinal microbiota. Recent scientific studies show an inverse correlation between the intake of flavonoids in the diet and the incidence of diabetes, such as to hypothesize the use of foods rich in flavonoids as potential food supplements in the management of diabetes. The cocoa flavonoids can bring benefits to the insulin-resistance condition by improving endothelial function, modifying glucose metabolism and reducing oxidative stress, which is considered the main cause of insulin resistance. In healthy individuals and even in patients with moderate cardiovascular risk, regular intake of flavonoids improves levels of cardiovascular biomarkers, reducing serum LDL cholesterol concentrations and triglycerides and increasing HDL cholesterol concentrations. The flavonoids present in cocoa may also inhibit platelet aggregation by down-regulation of the cellular synthesis of eicosanoids. Chocolate is an effective alternative for increasing fiber intake at recommended levels; in addition, it reduces intestinal transit time by increasing peristaltic movements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-35 years old
* Able to sign an informed consent

Exclusion Criteria:

* Refuse to sign an informed consent
* Diagnosis of organic diseases, including neoplastic inflammatory or cardiovascular diseases
* Drugs able to influence the gastrointestinal tract or interfering with symptoms
* Pregnancy
* Presence of diseases with a prognosis inferior to a year
* Hypersensitivity to chocolate or its components

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Organoleptic assessment | 1 day
  All subjects (n=10, matched per gender) will undergo a subjective organoleptic assessment of dark chocolate, based on a standard semi-quantitative scale (ranging 1-5) and a quantitative visual analogue scale (VAS, ranging from 0 to 100 on a horizontal line), to evaluate the visual, auditory, olfactory, gustatory and tactile aspects.
Gastrointestinal motility | 1 day
  All subjects (n=10, matched per gender) will be assessed for gastrointestinal motility in fasting state to monitor gastric empting, gallbladder empting (ultrasound) and oro-cecal transit time (H 2 lactulose BT), at baseline and at 5 minutes intervals during the firsts 30 minutes, and at 15 minutes intervals during the remaining 90 minutes, for a total of 2 hours of observations.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, MD, PhD, Principal Investigator — Clinica Medica "A. Murri", DIMO - University of Bari
Locations (1):
- Department of Biomedical Sciences Human Oncology - Clinica Medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Latif R. Chocolate/cocoa and human health: a review. Neth J Med. 2013 Mar;71(2):63-8. PMID 23462053
- [Background] Shah SR, Alweis R, Najim NI, Dharani AM, Jangda MA, Shahid M, Kazi AN, Shah SA. Use of dark chocolate for diabetic patients: a review of the literature and current evidence. J Community Hosp Intern Med Perspect. 2017 Sep 19;7(4):218-221. doi: 10.1080/20009666.2017.1361293. eCollection 2017 Oct. PMID 29181133
- [Background] Schroeter H, Heiss C, Balzer J, Kleinbongard P, Keen CL, Hollenberg NK, Sies H, Kwik-Uribe C, Schmitz HH, Kelm M. (-)-Epicatechin mediates beneficial effects of flavanol-rich cocoa on vascular function in humans. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):1024-9. doi: 10.1073/pnas.0510168103. Epub 2006 Jan 17. PMID 16418281
- [Background] Ueshima K. Magnesium and ischemic heart disease: a review of epidemiological, experimental, and clinical evidences. Magnes Res. 2005 Dec;18(4):275-84. PMID 16548143
- [Background] Allen RR, Carson L, Kwik-Uribe C, Evans EM, Erdman JW Jr. Daily consumption of a dark chocolate containing flavanols and added sterol esters affects cardiovascular risk factors in a normotensive population with elevated cholesterol. J Nutr. 2008 Apr;138(4):725-31. doi: 10.1093/jn/138.4.725. PMID 18356327
- [Background] Hayek N. Chocolate, gut microbiota, and human health. Front Pharmacol. 2013 Feb 7;4:11. doi: 10.3389/fphar.2013.00011. eCollection 2013. No abstract available. PMID 23405053
- [Background] Davinelli S, Corbi G, Righetti S, Sears B, Olarte HH, Grassi D, Scapagnini G. Cardioprotection by Cocoa Polyphenols and omega-3 Fatty Acids: A Disease-Prevention Perspective on Aging-Associated Cardiovascular Risk. J Med Food. 2018 Oct;21(10):1060-1069. doi: 10.1089/jmf.2018.0002. Epub 2018 May 3. PMID 29723102
- [Background] Mushref MA, Srinivasan S. Effect of high fat-diet and obesity on gastrointestinal motility. Ann Transl Med. 2013 Jul 1;1(2):14. doi: 10.3978/j.issn.2305-5839.2012.11.01. PMID 24432301
- [Background] Di Ciaula A, Wang DQ, Portincasa P. Gallbladder and gastric motility in obese newborns, pre-adolescents and adults. J Gastroenterol Hepatol. 2012 Aug;27(8):1298-305. doi: 10.1111/j.1440-1746.2012.07149.x. PMID 22497555